CLINICAL TRIAL: NCT04285385
Title: Aromatherapy With Lavender Essential Oil as a Complementary Treatment for the Control of Dental Anxiety in Patients Requiring Third Molar Surgery of the "University Autonomus Benito Juarez of Oaxaca" UABJO School of Dentistry
Brief Title: Aromatherapy With Lavender Essential Oil as a Complementary Treatment for the Control of Dental Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Autónoma Benito Juárez de Oaxaca (Other)
Responsible Party: Principal Investigator, Liliana Argueta Figueroa, Principal Investigator, Universidad Autónoma Benito Juárez de Oaxaca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19PEC001FO
Record Dates: First submitted 2020-02-21; First posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Dental Anxiety
Keywords: aromatherapy; lavender; anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aromatherapy (Experimental): 0.10 ml of lavender essential oil 30 minutes prior surgery
  Interventions: Other: Lavender aromatherapy
- Sham Aromatherapy (Sham Comparator): 0.10 ml mineral oil 30 minutes prior surgery
  Interventions: Other: Sham aromatherapy

INTERVENTIONS:
Other: Lavender aromatherapy — 0.10 ml of lavender essential oil
  Arms: Aromatherapy
Other: Sham aromatherapy — 0.10 ml of mineral oil
  Arms: Sham Aromatherapy

SUMMARY:
Dental anxiety is a common problem in dental care, the aim of this protocol is to evaluate the effect of lavender for the control of anxiety during a surgical dental extraction.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to take part in the study
* Healthy patients
* Patients signing the informed consent
* Patients who need surgical removal of third molars

Exclusion Criteria:

* Hypertensive patients
* Patients with nasal congestion problems
* Patients allergic to lavender.
* Patients under treatment with anti depressants

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Corah | 45 minutes before dental treatment
  Corah's Dental Anxiety Scale (1-25). Non anxiety (0-8), moderate (9-12), high (13-14), severe (over 15)
Cortisol | 5 minutes Before aromatherapy
  Salivary Cortisol Testing (ng/mL)
Cortisol | 30 minutes after aromatherapy
  Salivary Cortisol Testing (ng/mL)

SECONDARY OUTCOMES:
Heart rate | 5 minutes Before aromatherapy
  The speed of the heartbeat measured by the number of contractions of the heart per minute
Heart rate | 30 minutes after aromatherapy
  The speed of the heartbeat measured by the number of contractions of the heart per minute
Respiratory rate | 5 minutes Before aromatherapy
  The number of breaths per minute.
Respiratory rate | 30 minutes after aromatherapy
  The number of breaths per minute.
Arterial pressure | 5 minutes Before aromatherapy
  The pressure of circulating blood on the walls of blood vessels. (mm/Hg) sphingomanometer OMRON model HEM-7114
Arterial pressure | 30 minutes after aromatherapy
  The pressure of circulating blood on the walls of blood vessels. (mm/Hg) sphingomanometer OMRON model HEM-7114

CONTACTS AND LOCATIONS:
Overall Officials: Liliana Argueta-Figueroa, DMD PhD, Principal Investigator — UABJO

IPD SHARING:
Plan to Share IPD: Yes
Measures of cortisol, vital sign, Corah scale, sex and age.
Supporting Information: Study Protocol, ICF
Time Frame: Starting 6 months after publication in journal
Access Criteria: For meta analysis purposes, after contact with the PI